CLINICAL TRIAL: NCT00318565
Title: Navistar Thermocool Evaluation of the Catheter With the Stockert 70 Radiofrequency Generator for Endocardial Ablation in Patients With Typical Atrial Flutter
Brief Title: Catheter Evaluation for Endocardial Ablation in Patients With Typical Atrial Flutter
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BWI30031
Record Dates: First submitted 2006-04-25; First posted 2006-04-27 (Estimated); Results first posted 2010-03-02 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Atrial Flutter
Keywords: Heart Disease; Atrial Flutter; Typical Atrial Flutter
MeSH Terms: conditions — Atrial Flutter; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Navistar ThermoCool Catheter (Experimental)
  Interventions: Device: RF energy delivery for treatment of Typical Atrial flutter

INTERVENTIONS:
Device: RF energy delivery for treatment of Typical Atrial flutter — Navistar ThermoCool catheter
  Other Names: Therapeutic Catheters

SUMMARY:
The primary objective is to provide additional corroborative safety and efficacy data for the Navistar Thermocool catheter for the treatment of subjects with typical atrial flutter (AFL).

DETAILED DESCRIPTION:
This study is a prospective, non-randomized, single-arm, multi-center condition of approval evaluation. The device is currently FDA approved for commercial distribution. Subjects with symptomatic typical atrial flutter will be considered for the condition of approval study. This study will be conducted at up to 30 centers in a minimum of 221 evaluable subjects.

ELIGIBILITY:
Inclusion Criteria:

* Two symptomatic episodes of typical atrial flutter (or chronic atrial flutter) during the one-year period prior to enrollment. This may include typical AFL occurring while receiving anti-arrhythmic drug (AAD) therapy for non-AFL tachyarrhythmia, including atrial fibrillation.
* At least one episode of typical (clockwise or counterclockwise) atrial flutter documented by 12 lead electrocardiogram (ECG), Holter monitor, transtelephonic event monitor, telemetry strip, or implanted device within 6 months prior to enrollment.
* 18 years of age or older
* Informed consent

Exclusion Criteria:

* Intracardiac thrombus
* Uncontrolled heart failure, or New York Heart Association (NYHA) class III or IV heart failure
* Women who are pregnant
* Cardiac surgery (ventriculotomy or atriotomy) within the past two months
* Intra-atrial thrombus, tumor, or other abnormality that precludes catheter introduction and placement
* Unstable angina or acute myocardial infarction within 3 months
* Awaiting cardiac transplantation
* Heart disease in which corrective surgery is anticipated within 6 months
* Presence of condition that precludes appropriate vascular access
* Enrolled in any investigational device exemption (IDE) investigating study for a device or drug
* High risk for non-compliance with the protocol (e.g., inaccessible for follow-up by the investigator or patient's physician)
* Radio frequency (RF) ablation for typical atrial flutter within the past 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2006-01; Primary Completion 2007-09 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Warren Jackman, M.D., Principal Investigator — University of Oklahoma
Locations (23):
- United States (23):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Arizona Arrhythmia Consultants, Scottsdale, Arizona
  - Good Samaritan Hospital, Los Angeles, California
  - Pacific Heart Institute, Santa Monica, California
  - University of Florida, Gainsville, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - Florida Hospital, Orlando, Florida
  - University of Chicago, Chicago, Illinois
  - The Care Group LLC, St. Vincent Hospital and Health Care Center, Inc., Indianapolis, Indiana
  - Central Baptist Hospital, Lexington, Kentucky
  - Maine Medical Center, Portland, Maine
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Park Nicollet Institute, Minneapolis, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - University of Oklahoma, Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Heart Institute, Houston, Texas
  - University of Vermont, College of Medicine, Burlington, Vermont
  - INOVA Research Center, Falls Church, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrollment on June 7, 2006 Last subject enrolled August 14, 2007. Enrollment rate was 20.5 subjects per month across 21 hospitals
Groups:
- Ablation Group: Subjects to undergo ablation with the NaviStar ThermoCool catheter for the treatment of typical atrial flutter.
Period: Overall Study
Arm/Group | Ablation Group
Started | 291
Completed | 267
Not Completed | 24
Not completed — Excluded per protocol | 24

BASELINE CHARACTERISTICS:
Arm/Group | Ablation Group
Number analyzed (Participants) | 291
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 136
  >=65 years | 155
Age Continuous [Mean (Standard Deviation); unit: years] | 65.2 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 243
Region of Enrollment [Number; unit: participants]
  United States | 291

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Complete Bidirectional Conduction Block.
Description: Acute success is defined as the confirmation of complete bidirectional conduction block across the subeustachian (cavo-tricuspid) isthmus. The percentage of subjects with confirmed conduction block will serve as the outcome measure.
Time Frame: During the procedure
Population: Per protocol analysis. Number differs from "Participant Flow" because only 253 subjects were considered for the efficacy cohort.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ablation Group
Number analyzed (Participants) | 253
percentage of participants | 93.3 [90.1 to 100]
Statistical Analysis 1: Comparison: Ablation Group; An acute success rate of 88% is anticipated and the one-sided 95% lower confidence bound will be compared to 80%. The statistical hypothesis for the primary efficacy endpoint is evaluated as a one-tailed hypothesis at a = 0.05; Test type: Superiority or Other; p = .05, Exact binomial distribution; Binomial distribution = 93.3, 95% CI 1-sided [lower limit 90.1]

2. Primary Outcome: Percentage of Subjects Experiencing Cardiovascular Specific Adverse Events (CSAE) Within Seven (7) Days of the Ablation Procedure.
Description: The cardiovascular specific adverse event (CSAE) rate is the primary safety enpoint for the study. A CSAE is an event which occurs within the first week (7 days) following use of the device and is one of the following cardiac specific adverse events: cardiac perforation, pericardial effusion, pulmonary embolus, complete heart block, stroke, acute myocardial infarction, and death.
Time Frame: 7 Days
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ablation Group
Number analyzed (Participants) | 267
percentage of participants | 1.5 [0 to 3.4]
Statistical Analysis 1: Comparison: Ablation Group; The anticipated rate of the CSAE is 2.7% and the one-sided 95% upper confidence bound will be compared to 7%; Test type: Superiority or Other; p = .05, Exact Binomial Distribution; Binomial Distribution = 1.5, 95% CI 1-sided [upper limit 7]

ADVERSE EVENTS:
Arm/Group | Ablation Group
Serious Adverse Events (participants affected / at risk) | 4/267
Other Adverse Events (participants affected / at risk) | 73/267
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ablation Group (N=267)
Pulmonary Embolus (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Complete Heart Block (Cardiac disorders) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ablation Group (N=267)
Adverse Events within 7 Days- Device Related (General disorders) | 1 (1)
Adverse Events within 7 Days- Possibly Device Related (General disorders) | 0 (0)
Adverse Events within 7 Days- Procedure Related (General disorders) | 18 (21)
Adverse Events within 7 Days- Possibly Procedure Related (General disorders) | 12 (12)
Adverse Events within 7 Days- Unrelated to Device or Procedure (General disorders) | 24 (29)
Adverse Events Greater than 7 Days- Device Related (General disorders) | 0 (0)
Adverse Events Greater than 7 Days- Possibly Device Related (General disorders) | 0 (0)
Adverse Events Greater than 7 Days- Procedure Related (General disorders) | 2 (2)
Adverse Events Greater than 7 Days- Possibly Procedure Related (General disorders) | 0 (0)
Adverse Events Greater than 7 Days- Unrelated to Device or Procedure (General disorders) | 28 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No